CLINICAL TRIAL: NCT02660580
Title: A Randomized, Double-blind Trial to Evaluate the Efficacy, Safety and Immunogenicity of MSB11022 Compared With Humira® in Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: MSB11022 in Moderate to Severe Chronic Plaque Psoriasis
Acronym: AURIEL-PsO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fresenius Kabi SwissBioSim GmbH (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR200588-002; 2015-003287-37 (EudraCT Number)
Record Dates: First submitted 2016-01-17; First posted 2016-01-21 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Psoriasis; Plaque Type Psoriasis; Moderate to Severe Plaque Psoriasis
Keywords: Adalimumab; MSB11022; Psoriasis; Phase III
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MSB11022 (Core Treatment Period) (Experimental): Participants received MSB11022 subcutaneously at an initial dose of 80 milligram (mg) on Day 1 of Week 1 followed by 40 mg every other week starting at Week 2 up to and including Week 14 in Core Treatment Period.
  Interventions: Drug: MSB11022
- EU-Humira (Active Comparator): Participants received EU-Humira subcutaneously at an initial dose of 80 mg on Day 1 of Week 1 followed by 40 mg every other week starting at Week 2 up to and including Week 14 in Core Treatment Period.
  Interventions: Drug: Humira®
- MSB11022 (Extended Treatment Period) (Experimental): Participants who had achieved PASI 50 and received MSB11022 during Core Treatment Period continued to receive MSB11022 subcutaneously at dose of 40 mg every other week starting at Week 16 up to and including Week 50 in extended treatment period.
  Interventions: Drug: MSB11022
- EU-Humira/EU-Humira (Active Comparator): Participants who had achieved PASI 50 and received EU-Humira in Core Treatment Period and continued to receive EU-Humira subcutaneously at dose of 40 mg every other week starting at Week 16 up to and including Week 50 after re-randomization in extended treatment period.
  Interventions: Drug: Humira®
- EU-Humira/MSB11022 (Experimental): Participants who had achieved PASI 50 and received EU-Humira in Core Treatment Period were re-randomized to receive MSB11022 subcutaneously at dose of 40 mg every other week starting at Week 16 up to and including Week 50 in extended treatment period.
  Interventions: Drug: MSB11022; Drug: Humira®

INTERVENTIONS:
Drug: MSB11022 — Participants received MSB11022 drug subcutaneously MSB11022 (Core Treatment Period), MSB11022 (Extended Treatment Period) and EU-Humira/MSB11022 arm.
  Arms: EU-Humira/MSB11022; MSB11022 (Core Treatment Period); MSB11022 (Extended Treatment Period)
Drug: Humira® — Participants received EU-Humira subcutaneously in EU-Humira, EU-Humira/EU-Humira and EU-Humira/MSB11022 arm.
  Arms: EU-Humira; EU-Humira/EU-Humira; EU-Humira/MSB11022

SUMMARY:
The purpose of this study was to compare the efficacy, safety and immunogenicity of MSB11022 and Humira® in adult subjects with moderate to severe chronic plaque type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants greater than or equal to (>=) 18 years old with a clinical diagnosis of stable moderate to severe plaque psoriasis (defined by Psoriasis Area and Severity Index [PASI] score >=12, Physician Global Assessment [PGA] score >=3, and >=10% of body surface area affected at Screening and Baseline [Day 1 of Week 1]) who have a history of receipt of or are candidates for systemic therapy or phototherapy for active plaque-type psoriasis despite topical therapy
* Participants must not have received more than 1 biologic therapy
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Participants was excluded if they have erythrodermic, pustular, guttate, or medication-induced forms of psoriasis or other active skin diseases/infections that may interfere with the evaluation of plaque psoriasis
* Participants must not have received adalimumab or an investigational or licensed biosimilar of adalimumab; topical therapies for the treatment of psoriasis or ultraviolet B phototherapy within 2 weeks of investigational medicinal product (IMP) administration or plan to take such treatment during the trial; or psoralen combined with ultraviolet A phototherapy or nonbiological systemic therapies for psoriasis within 4 weeks prior to IMP administration
* Participants was excluded if they have a history of an ongoing, chronic, or recurrent infectious disease (except for latent tuberculosis [TB]); history of active TB; or a history of hypersensitivity to any component of the IMP formulation, comparable drugs, or latex
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Fresenius Kabi Swiss BioSim GmbH
Locations (76):
- United States (6):
  - San Luis Dermatology & Laser Clinic, Inc., San Luis Obispo, California
  - Florida Academic Centers Research and Education, Coral Gables, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Modern Research Associates, Dallas, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
- Bulgaria (11):
  - DCC 'Sveti Georgi' EOOD, Haskovo
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - DCC "Sv. Georgi", EOOD, Plovdiv
  - Diagnostic Consultative Center II - Sofia OOD, Sofia
  - MC "Robert Koch", EOOD, Sofia
  - Medical Center "Excelsior", OOD, Sofia
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - DCC 3 - Varna, EOOD, Varna
- Canada (9):
  - Stratica Medical, Edmonton, Alberta
  - Dr. Lorne E. Albrecht, Inc., Surrey, British Columbia
  - Gupta, Aditya K. MD, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - Dr Melinda Gooderham Medicine Professional Corporation, Peterborough, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Centre de Recherche Dermatologique du Quebec Metropolitain, Ste-Foy, Quebec
- Czechia (7):
  - Nemocnice Jihlava, Jihlava
  - Nemocnice Novy Jicin a.s., Nový Jičín
  - Fakultni nemocnice Olomouc, Olomouc
  - Clintrial, s.r.o., Prague
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Dermatovenerologická klinika, Praha 8 - Liben
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- Estonia (4):
  - Vahlberg & Pild OÜ, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - Clinical Research Centre, Tartu
  - Tartu University Hospital, Tartu
- France (4):
  - CHU Nice - Hôpital de l'Archet 2, Nice, Alpes Maritimes
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Maison du Haut Lévêque, Bordeaux, Gironde
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Hôpital de la Timone, Marseille
- Germany (5):
  - Licca, Augsburg, Bavaria
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia
  - Praxis fuer Dermatologie und Venerologie, Dresden, Saxony
  - Clinical Research Hamburg GmbH, Hamburg
- Hungary (5):
  - Ambrozia Gondozohaz Szolg. Nonprofit Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - ALLERGO-DERM BAKOS Kft., Szolnok
- Mexico (7):
  - Clinica de Investigacion en Reumatologia y Obesidad S.C., Guadalajara, Jalisco
  - Unidad de Investigacion de las Enfermedades Reumaticas, Cuauhtémoc, Mexico City
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Clinical Research Institute S.C., Tlalnepantla, State of Mexico
  - Köhler & Milstein Research S.A de C.V., Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo Especializado de la Investigacion Clinica en Yucatan, Mérida, Yucatán
  - Derma Norte del Bajio S.C., Aguascalientes
- Poland (12):
  - Centrum Kliniczno - Badawcze J. Brzezicki, B. Górnikiewicz-Brzezicka Lekarze Spółka Partnerska, Elblag
  - Gdanskie Centrum Zdrowia Sp. z o.o., Gdansk
  - Centrum Medyczne Plejady, Krakow
  - Grazyna Pulka Specjalistyczny Osrodek "ALL-MED", Krakow
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska sp. komandytowo-akcyjna, Lodz
  - NZOZ ALL-MED Centrum Medyczne Specjalistyczne Gabinety Lekarskie, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej "Med-Laser", Lublin
  - Centrum Badan Klinicznych S.C., Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Niepubliczny Zaklad Opieki Zdrowotnej "Nasz Lekarz" Praktyka Grupowa Lekarzy Rodzinnych z, Torun
  - SP Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
  - Centrum Medyczne ADAMAR, Wroclaw
- Russia (4):
  - SBEI HPE "Kazan State Medical University" of the MoH of the RF, Kazan'
  - LLC "Alliance Biomedical - Russian Group", Saint Petersburg
  - Clinic of skin and veneral diseases, Saratov
  - SBEI HPE "Yaroslavl State Medical University" of the MoH of the RF, Yaroslavl
- United Kingdom (2):
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Russells Hall Hospital, Dudley, West Midlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to either MSB11022 or EU-Humira in Core Treatment Period till Week 16. Participants who achieved PASI50 at Week 16 entered Extension Period where participants in MSB11022 were continued to receive MSB11022 & participants in EU-Humira were re-randomized to receive either MSB11022 or EU-Humira for additional 37 weeks.
Period: Core Treatment Period (Week 1 to 16)
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Started | 222 | 221 | 0 | 0 | 0
Treated | 221 | 220 | 0 | 0 | 0
Completed | 213 | 202 | 0 | 0 | 0
Not Completed | 9 | 19 | 0 | 0 | 0
Not completed — Randomized, not treated | 1 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 1 | 0 | 0 | 0
Not completed — Other un-specified | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 9 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0 | 0
Period: Extended Treatment Period(Week 16 to 52)
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Started | 0 | 0 | 213 | 101 | 101
Completed | 0 | 0 | 195 | 90 | 90
Not Completed | 0 | 0 | 18 | 11 | 11
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 1
Not completed — Other un-specified | 0 | 0 | 1 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 4 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 8 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira | Total
Number analyzed (Participants) | 222 | 221 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.8) | 42.7 (12.0) | 43.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 73 | 148
  Male | 147 | 148 | 295
Race [Count of Participants; unit: Participants]
  White | 205 | 200 | 405
  Black or African American | 2 | 1 | 3
  Asian | 5 | 9 | 14
  American Indian or Alaska Native | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 1 | 1
  Missing/Not collected at this site | 0 | 2 | 2
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 23 | 46
  Not Hispanic or Latino | 199 | 196 | 395
  Missing | 0 | 2 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in PASI at Week 16
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72, with higher scores reflecting more disease severity. Percent change from Baseline in PASI score was reported.
Time Frame: Baseline (Day 1 of Core Treatment Period), Week 16
Population: The PP Analysis set was used.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Percent change | -90.6 (11.3) [lower limit 11.3] | -91.7 (9.9) [lower limit 9.9]
Statistical Analysis 1: Comparison: MSB11022 (Core Treatment Period) vs EU-Humira; Test type: Equivalence — MSB11022 was considered equivalent to EU-Humira if the 95% CI for the treatment difference was included in the equivalence interval [-15%, 15%]); Least Square (LS) Mean difference = 0.88, 95% CI 2-sided [-1.21 to 2.98]

2. Secondary Outcome: Percentage of Participants Who Achieved PASI 50, 90 and 100 at Week 16
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72 with higher scores reflecting more disease severity. The PASI 50, 90 and 100 response rate at Week 16 is measured as the percentage of participants who achieved at least 50, 90 and 100% improvement from baseline PASI score at Week 16.
Time Frame: Week 16
Population: PP analysis set was used.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Percentage of Participants
  PASI 50 | 100.0 | 100.0
  PASI 90 | 64.0 | 66.0
  PASI 100 | 33.0 | 37.2

3. Secondary Outcome: Percentage of Participants Who Achieved PASI 50, 75, 90 and 100 at Week 24
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72 with higher scores reflecting more disease severity. The PASI response rate at Week 24 is measured as the percentage of participants who achieved at least 50, 75, 90 and 100% improvement from baseline PASI at Week 24.
Time Frame: Week 24
Population: The Extended Treatment Period (ETP)-PP Analysis Set included participants who were in PP Analysis Set & were re-randomized & received treatment in Extended Treatment Period. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 200 | 94 | 92
Percentage of Participants
  PASI 50 | 100.0 | 98.9 | 100.0
  PASI 75 | 92.5 | 88.3 | 94.6
  PASI 90 | 74.0 | 78.7 | 80.4
  PASI 100 | 42.5 | 37.2 | 35.9

4. Secondary Outcome: Percentage of Participants Who Achieved PASI 50, 75, 90 and 100 at Week 52
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72 with higher scores reflecting more disease severity. The PASI response rate at Week 52 is measured as the percentage of participants who achieved at least 50, 75, 90 and 100% improvement from baseline PASI at Week 52.
Time Frame: Week 52
Population: The ETP-PP Analysis Set was used. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 186 | 85 | 87
Percentage of Participants
  PASI 50 | 97.8 | 100.0 | 100.0
  PASI 75 | 90.9 | 92.9 | 93.1
  PASI 90 | 76.3 | 78.8 | 85.1
  PASI 100 | 53.8 | 54.1 | 57.5

5. Secondary Outcome: Percent Change From Baseline in PASI at Week 24 and 52
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72, with higher scores reflecting more disease severity.
Time Frame: Baseline (Day 1 of Extended Treatment Period), Weeks 24 and 52
Population: The ETP-PP analysis set was used. Here "Number analyzed" Signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
Percent change
  Week 24: number analyzed (Participants) | 200 | 94 | 92
  Week 24 | -92.9 (9.9) | -91.3 (12.7) | -94.2 (8.2)
  Week 52: number analyzed (Participants) | 186 | 85 | 87
  Week 52 | -92.8 (13.6) | -93.9 (9.6) | -94.8 (9.7)

6. Secondary Outcome: Number of Participants With Change From Baseline in Physician's Global Assessment (PGA) Score to "Clear" or "Almost Clear" at Week 16
Description: PGA was assessed relative to baseline condition based on a scale ranged from 0 to 4, where 0 indicates Clear condition (no signs of psoriasis, post-inflammatory hyperpigmentation may be present), 1 indicates Almost clear condition (normal to pink coloration of lesion, no thickening and no to minimal [focal] scaling), 2 indicates Mild condition (pink to light red coloration, just detectable to mild thickening and predominantly fine scaling), 3 indicates Moderate condition (dull bright red, clearly distinguishable erythema, clearly distinguishable to moderate thickening and moderate scaling), and 4 indicates Severe condition (bright to deep dark red coloration, severe thickening with hard edges and severe/coarse scaling covering almost all or all lesions).
Time Frame: Baseline (Day 1 of Core Treatment Period), Week 16
Population: PP Analysis set was used. Number of participants with PGA response of Clear or Almost clear at Week 16 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Participants
  Baseline: Moderate; Week 16: Clear | 52 | 51
  Baseline: Moderate; Week 16: Almost clear | 76 | 59
  Baseline: Severe; Week 16: Clear | 16 | 20
  Baseline: Severe; Week 16: Almost clear | 27 | 26

7. Secondary Outcome: Number of Participants With Change From Baseline in Physician's Global Assessment (PGA) Score to "Clear" or "Almost Clear" at Week 24 and 52
Description: as for outcome 6
Time Frame: Baseline (Day 1 of Extended Treatment Period), Week 24 and 52
Population: ETP-PP Analysis set was used. Here "Number analyzed" indicates number of participants who were evaluable for this outcome measure at specified category. Number of participants with PGA response of Clear or Almost clear at Week 24 and 52 were presented.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
Participants
  Baseline: Moderate; Week 24: Clear: number analyzed (Participants) | 200 | 94 | 92
  Baseline: Moderate; Week 24: Clear | 69 | 25 | 25
  Baseline: Moderate; Week 24: AlmostClear: number analyzed (Participants) | 200 | 94 | 92
  Baseline: Moderate; Week 24: AlmostClear | 52 | 24 | 31
  Baseline: Severe; Week 24: Clear: number analyzed (Participants) | 200 | 94 | 92
  Baseline: Severe; Week 24: Clear | 18 | 11 | 9
  Baseline: Severe; Week 24: Almost Clear: number analyzed (Participants) | 200 | 94 | 92
  Baseline: Severe; Week 24: Almost Clear | 27 | 14 | 13
  Baseline: Moderate; Week 52: Clear: number analyzed (Participants) | 188 | 85 | 87
  Baseline: Moderate; Week 52: Clear | 74 | 29 | 34
  Baseline: Moderate; Week 52: AlmostClear: number analyzed (Participants) | 188 | 85 | 87
  Baseline: Moderate; Week 52: AlmostClear | 40 | 13 | 16
  Baseline: Severe; Week 52: Clear: number analyzed (Participants) | 188 | 85 | 87
  Baseline: Severe; Week 52: Clear | 29 | 17 | 16
  Baseline: Severe; Week 52: Almost Clear: number analyzed (Participants) | 188 | 85 | 87
  Baseline: Severe; Week 52: Almost Clear | 15 | 6 | 6

8. Secondary Outcome: Time to Achieve PASI 50
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72, with higher scores reflecting more disease severity. Time to achieve at least 50% improvement in PASI from baseline was measured.
Time Frame: Baseline (Day 1 of Core Treatment Period) up to Month 4
Population: PP analysis set was used.
Measure: Median (Full Range); unit: Months
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Months | 1.6 (0.2) [0.2 to 3.7] | 1.6 (0.2) [0.2 to 3.5]

9. Secondary Outcome: Time to Achieve PASI 75
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72, with higher scores reflecting more disease severity. Time to achieve at least 75% improvement in PASI from baseline was measured.
Time Frame: Baseline (Day 1 of Core Treatment Period) up to Month 4
Population: PP analysis set was used.
Measure: Median (Full Range); unit: Months
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Months | 2.5 (0.2) [0.2 to 3.5] | 1.7 (0.7) [0.7 to 3.7]

10. Secondary Outcome: Time to Achieve PASI 90
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72, with higher scores reflecting more disease severity. Time to achieve at least 90% improvement in PASI from baseline was measured.
Time Frame: Baseline (Day 1 of Core Treatment Period) up to Month 4
Population: PP analysis set was used.
Measure: Median (Full Range); unit: Months
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Months | 3.4 (0.7) [0.7 to 3.5] | 2.6 (1.4) [1.4 to 3.7]

11. Secondary Outcome: Time to Achieve PASI 100
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72, with higher scores reflecting more disease severity. Time to achieve at least 100% improvement in PASI from baseline was measured.
Time Frame: Baseline (Day 1 of Core Treatment Period) up to Month 13.5
Population: ETP-PP analysis set was used.
Measure: Median (Full Range); unit: Month
Groups:
- MSB11022 (Overall Treatment Period): Participants received MSB11022 subcutaneously at dose of 40 mg every other week starting at Week 1 up to and including Week 50 in overall treatment period.
- EU-Humira/EU-Humira (Overall Treatment Period): Participants who received EU-Humira up to Week 16 continued to receive EU-Humira subcutaneously at dose of 40 mg every other week starting at Week 16 up to and including Week 50 after re-randomization in overall treatment period.
- EU-Humira/MSB11022 (Overall Treatment Period): Participants who received EU-Humira up to Week 16 were re-randomized to receive MSB11022 subcutaneously at dose of 40 mg every other week starting at Week 16 up to and including Week 50 in overall treatment period.
Arm/Group | MSB11022 (Overall Treatment Period) | EU-Humira/EU-Humira (Overall Treatment Period) | EU-Humira/MSB11022 (Overall Treatment Period)
Number analyzed (Participants) | 203 | 95 | 96
Month | 7.2 [0.7 to 11.8] | 7.2 [1.6 to 11.8] | 8.9 [1.6 to 11.8]

12. Secondary Outcome: Number of Participants With Change in Physician's Global Assessment (PGA) From Baseline at Week 16
Description: as for outcome 6
Time Frame: Baseline (Day 1 of Core Treatment Period), Week 16
Population: PP Analysis set was used. Only categories for which participants recorded a PGA response were included below.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Participants
  Baseline- Moderate; Week 16- Clear | 52 | 51
  Baseline- Moderate; Week 16- Almost Clear | 76 | 59
  Baseline- Moderate; Week 16- Mild | 16 | 17
  Baseline- Moderate; Week 16- Moderate | 2 | 1
  Baseline- Severe; Week 16- Clear | 16 | 20
  Baseline- Severe; Week 16- Almost Clear | 27 | 26
  Baseline- Severe; Week 16- Mild | 12 | 16
  Baseline- Severe; Week 16- Moderate | 2 | 1

13. Secondary Outcome: Number of Participants With Change in Physician's Global Assessment (PGA) From Baseline at Week 24
Description: as for outcome 6
Time Frame: Baseline (Day 1 of Extended Treatment Period), Week 24
Population: ETP-PP Analysis set was used. Only categories for which participants recorded a PGA response were included below. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 200 | 94 | 92
Participants
  Baseline- Moderate; Week 24- Clear | 69 | 25 | 25
  Baseline- Moderate; Week 24- Almost Clear | 52 | 24 | 31
  Baseline- Moderate; Week 24- Mild | 21 | 10 | 7
  Baseline- Moderate; Week 24- Moderate | 2 | 2 | 0
  Baseline- Severe; Week 24- Clear | 18 | 11 | 9
  Baseline- Severe; Week 24- Almost Clear | 27 | 14 | 13
  Baseline- Severe; Week 24- Mild | 9 | 6 | 6
  Baseline- Severe; Week 24- Moderate | 2 | 1 | 1
  Baseline- Severe; Week 24- Severe | 0 | 1 | 0

14. Secondary Outcome: Number of Participants With Change in Physician's Global Assessment (PGA) From Baseline at Week 52
Description: as for outcome 6
Time Frame: Baseline (Day 1 of Extended Treatment Period), Week 52
Population: ETP-PP Analysis set was used. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure. Only categories for which participants recorded a PGA response were included below.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 188 | 85 | 87
Participants
  Baseline- Moderate; Week 52- Clear | 74 | 29 | 34
  Baseline- Moderate; Week 52- Almost Clear | 40 | 13 | 16
  Baseline- Moderate; Week 52- Mild | 17 | 11 | 6
  Baseline- Moderate; Week 52- Moderate | 4 | 0 | 4
  Baseline- Moderate; Week 52- Missing | 1 | 0 | 0
  Baseline- Severe; Week 52- Clear | 29 | 17 | 16
  Baseline- Severe; Week 52- Almost Clear | 15 | 6 | 6
  Baseline- Severe; Week 52- Mild | 3 | 7 | 3
  Baseline- Severe; Week 52- Moderate | 3 | 2 | 2
  Baseline- Severe; Week 52- Severe | 1 | 0 | 0
  Baseline- Severe; Week 52- Missing | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs of Special Interest and TEAEs Leading to Death up to Week 16
Description: Adverse event(AE) was defined as any untoward medical occurrence in participants which does not necessarily have causal relationship with treatment. AE was any unfavorable and unintended sign(including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. A serious adverse event(SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline (Day 1 of Core Treatment Period) up to Week 16
Population: Safety (SAF) Analysis Set included all randomized participants who received at least 1 dose of MSB11022 or EU-Humira. Participants in SAF were analyzed according to actual treatment received initially during the relevant treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 221 | 220
Participants
  Participants with TEAEs | 114 | 117
  Participants with Serious TEAEs | 8 | 6
  Participants with TEAEs of special interest | 2 | 3
  Participants with TEAEs Leading to Death | 0 | 0

16. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs of Special Interest and TEAEs Leading to Death up to Week 54
Description: as for outcome 15
Time Frame: Baseline (Day 1 of Extended Treatment Period) up to Week 54
Population: ETP-SAF Analysis Set was used. Participants were analyzed according to actual treatment received initially during the relevant treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 213 | 101 | 101
Participants
  Participants with TEAEs | 142 | 65 | 63
  Participants with Serious TEAEs | 12 | 3 | 4
  Participants with TEAEs of special interest | 10 | 1 | 4
  Participants with TEAEs Leading to Death | 0 | 1 | 0

17. Primary Outcome: Percentage of Participants Who Achieved Psoriasis Area and Severity Index 75 (PASI 75) at Week 16
Description: PASI correlates to the physician's assessment of psoriasis symptoms including redness of lesions, thickness of lesions, scaliness of lesions and extent of disease. Each parameter is graded from 0-4, 0 refers to no disease and 4 to severe involvement. The body is divided into 4 areas for scoring (head, arms, trunk to groin, legs to top of buttocks), and the final score ranges from 0-72 with higher scores reflecting more disease severity. The PASI-75 response is defined as the percentage of participants who achieved at least a 75% improvement in PASI score from Baseline.
Time Frame: Week 16
Population: The per-protocol (PP) Analysis Set included all randomized and treated participants who did not have any major protocol deviations during the Core Treatment Period with respect to factors likely to affect the efficacy of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Percentage of Participants | 89.7 | 91.6
Statistical Analysis 1: Comparison: MSB11022 (Core Treatment Period) vs EU-Humira; Test type: Equivalence — MSB11022 was considered equivalent to EU-Humira if the 95% stratified Newcombe Confidence Interval (CI) for the difference in percentage was included in the equivalence interval (-18, 18); Percentage difference = -1.9, 95% CI 2-sided [-7.82 to 4.07]

18. Secondary Outcome: Number of Participants With Clinically Meaningful Differences in Laboratory Values
Description: Based on categories of low, normal, or high according to the laboratory normal ranges, there were no clinically meaningful differences across the treatment groups in the numbers of participants with shifts in Laboratory parameters including hematology, chemistry and urinalysis from normal at Core Baseline to either low or high during the overall treatment period. Clinical meaningful was determined by the investigator.
Time Frame: Core Treatment Period: Baseline up to 16; Extended Treatment Period: Baseline up to Week 54
Population: Safety Analysis Set (SAF) was used for up to Week 16. The ETP-SAF was used in Extended Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | MSB11022 (Extended Treatment Period) | EU-Humira | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 221 | 213 | 220 | 101 | 101
Participants | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Anti-nuclear Antibodies (ANA) and Anti-double-stranded Deoxyribonucleic Acid (Anti-dsDNA) Assessments at Week 16
Description: Number of participants ANA and anti-ds DNA values were reported. For ANA, positivity is defined as any participants with ANA titer greater than (>) 1:160 and negativity is defined as ANA titer less than (<) 1:160. For anti-ds DNA, positivity is defined as any participants with adsDNA > 15 units per milliliter (U/mL), intermediate category is defined as value between 10 U/mL to 15 U/mL and negativity is defined as adsDNA < 10 U/mL.
Time Frame: Week 16
Population: Safety analysis set was used.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 221 | 220
Participants
  Participants with Negative ANA values | 205 | 190
  Participants with Positive ANA values | 6 | 10
  Participants with Negative anti-ds DNA values | 201 | 186
  Participants with Intermediate anti-ds DNA values | 4 | 5
  Participants with Positive anti-ds DNA values | 4 | 6

20. Secondary Outcome: Number of Participants With Anti-nuclear Antibodies (ANA) and Anti-double-stranded Deoxyribonucleic Acid (Anti-dsDNA) Assessments at Week 24, 32, 40 and 52
Description: as for outcome 19
Time Frame: Week 24, 32, 40 and 52
Population: ETP-SAF included all re-randomized participants who received at least 1 dose of MSB11022 or EU-approved Humira in ETP. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure & "Number analyzed" signifies those participants who were evaluable for this outcome measure for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 213 | 101 | 101
Participants
  Week 24: Negative ANA: number analyzed (Participants) | 201 | 94 | 97
  Week 24: Negative ANA | 188 | 89 | 92
  Week 32: Negative ANA: number analyzed (Participants) | 199 | 88 | 95
  Week 32: Negative ANA | 186 | 85 | 88
  Week 40: Negative ANA: number analyzed (Participants) | 196 | 91 | 92
  Week 40: Negative ANA | 178 | 85 | 85
  Week 52: Negative ANA: number analyzed (Participants) | 193 | 87 | 87
  Week 52: Negative ANA | 185 | 84 | 79
  Week 24: Positive ANA: number analyzed (Participants) | 201 | 94 | 97
  Week 24: Positive ANA | 13 | 5 | 5
  Week 32: Positive ANA: number analyzed (Participants) | 199 | 88 | 95
  Week 32: Positive ANA | 13 | 3 | 7
  Week 40: Positive ANA: number analyzed (Participants) | 196 | 91 | 92
  Week 40: Positive ANA | 18 | 6 | 7
  Week 52: Positive ANA: number analyzed (Participants) | 193 | 87 | 87
  Week 52: Positive ANA | 8 | 3 | 8
  Week 24: Negative anti-dsDNA: number analyzed (Participants) | 202 | 95 | 94
  Week 24: Negative anti-dsDNA | 191 | 89 | 88
  Week 32: Negative anti-dsDNA: number analyzed (Participants) | 199 | 88 | 93
  Week 32: Negative anti-dsDNA | 184 | 83 | 86
  Week 40: Negative anti-dsDNA: number analyzed (Participants) | 196 | 91 | 92
  Week 40: Negative anti-dsDNA | 179 | 86 | 84
  Week 52: Negative anti-dsDNA: number analyzed (Participants) | 192 | 87 | 88
  Week 52: Negative anti-dsDNA | 173 | 81 | 79
  Week 24: Positive anti-dsDNA: number analyzed (Participants) | 202 | 95 | 94
  Week 24: Positive anti-dsDNA | 8 | 3 | 5
  Week 32: Positive anti-dsDNA: number analyzed (Participants) | 199 | 88 | 93
  Week 32: Positive anti-dsDNA | 8 | 3 | 5
  Week 40: Positive anti-dsDNA: number analyzed (Participants) | 196 | 91 | 92
  Week 40: Positive anti-dsDNA | 10 | 3 | 7
  Week 52: Positive anti-dsDNA: number analyzed (Participants) | 192 | 87 | 88
  Week 52: Positive anti-dsDNA | 11 | 2 | 7
  Week 24: Intermediate anti-dsDNA: number analyzed (Participants) | 202 | 95 | 94
  Week 24: Intermediate anti-dsDNA | 3 | 3 | 1
  Week 32: Intermediate anti-dsDNA: number analyzed (Participants) | 199 | 88 | 93
  Week 32: Intermediate anti-dsDNA | 7 | 2 | 2
  Week 40: Intermediate anti-dsDNA: number analyzed (Participants) | 196 | 91 | 92
  Week 40: Intermediate anti-dsDNA | 7 | 2 | 1
  Week 52: Intermediate anti-dsDNA: number analyzed (Participants) | 192 | 87 | 88
  Week 52: Intermediate anti-dsDNA | 8 | 4 | 2

21. Secondary Outcome: Number of Participants With Clinically Meaningful Differences in Vital Signs
Description: Number of participants with clinically meaningful abnormalities in vital signs were reported. Clinical meaningful was determined by the investigator.
Time Frame: Core Treatment Period: Baseline up to 16; Extended Treatment Period: Baseline up to Week 54
Population: Safety analysis set was used for Core Treatment Period. ETP-SAF was used for Extended Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | MSB11022 (Extended Treatment Period) | EU-Humira | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 221 | 213 | 220 | 101 | 101
Participants | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in 12-Electrocardiogram (12-ECG)
Description: Number of participants with clinically significant abnormalities in 12-ECG were reported. Clinical significance was determined by the investigator.
Time Frame: Core Treatment Period: Baseline up to 16; Extended Treatment Period: Baseline up to Week 54
Population: Safety analysis set was used for Core Treatment Period. ETP-SAF was used for Extended Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | MSB11022 (Extended Treatment Period) | EU-Humira | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 221 | 213 | 220 | 101 | 101
Participants | 0 | 1 | 0 | 1 | 1

23. Secondary Outcome: Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item validated quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The DLQI measures how much participant's skin problems has affected his life. Responses range from 0=Not at all to 3=Very much. The DLQI total score is the sum of individual 10 items and could range from 0 to 30 (higher score indicated greater negative impact on life).
Time Frame: Weeks 16
Population: PP analysis set was used.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 203 | 191
Units on a scale | 2.4 (3.2) [lower limit 3.2] | 2.5 (3.7) [lower limit 3.7]

24. Secondary Outcome: Dermatology Life Quality Index (DLQI) at Week 24 and 52
Description: as for outcome 23
Time Frame: Week 24 and 52
Population: ETP-PP analysis set was used. Here "Number analyzed" signifies number of participants who were evaluable for this outcome measure at specified category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
Units on a scale
  Week 24: number analyzed (Participants) | 200 | 94 | 92
  Week 24 | 2.5 (4.1) | 2.3 (4.0) | 2.3 (3.9)
  Week 52: number analyzed (Participants) | 186 | 85 | 86
  Week 52 | 3.0 (4.7) | 2.1 (3.5) | 2.7 (4.0)

25. Secondary Outcome: European Quality of Life 5-Dimensions and 5-Levels Questionnaire (EQ5D-5L) Descriptive Score at Week 16
Description: The EQ-5D-5L questionnaire assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The participant was asked to indicate his/her current health state by selecting the most appropriate level in each of the 5 dimensions. The responses are converted into a single index value, with scores ranging from -0.594 to 1 (a higher score indicates better health state).
Time Frame: Week 16
Population: PP analysis set was used. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 189 | 179
Units on a scale | 0.9 (0.1) [lower limit 0.1] | 0.9 (0.1) [lower limit 0.1]

26. Secondary Outcome: European Quality of Life 5-Dimensions and 5-Levels Questionnaire (EQ5D-5L) Descriptive Score at Week 24 and 52
Description: as for outcome 25
Time Frame: Week 24 and 52
Population: ETP-PP analysis set was used. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified category.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
Units on a scale
  Week 24: number analyzed (Participants) | 200 | 94 | 92
  Week 24 | 0.8 (0.1) | 0.9 (0.1) | 0.9 (0.1)
  Week 52: number analyzed (Participants) | 186 | 85 | 86
  Week 52 | 0.9 (0.1) | 0.9 (0.1) | 0.8 (0.1)

27. Secondary Outcome: European Quality of Life 5-Dimensions and 5-Levels Questionnaire (EQ5D-5L) Based on Visual Analogue Scale (VAS) Score at Week 16
Description: The EQ-5D-5L questionnaire assesses 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response options (no problems, slight problems, moderate problems, severe problems and extreme problems) that reflect increasing levels of difficulty. The participant was asked to indicate his/her current health state by selecting the most appropriate level on a visual analog scale, where the participant was asked to rate current health status on a scale of 0 to 100, with 0 being the worst imaginable health state.
Time Frame: Week 16
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 189 | 179
Units on a scale | 81.9 (13.9) [lower limit 13.9] | 83.1 (15.0) [lower limit 15.0]

28. Secondary Outcome: European Quality of Life 5-Dimensions and 5-Levels Questionnaire (EQ5D-5L) Based on VAS Score at Week 24 and 52
Description: as for outcome 27
Time Frame: Week 24 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
Units on a scale
  Week 24: number analyzed (Participants) | 200 | 94 | 92
  Week 24 | 83.2 (14.2) | 84.2 (13.7) | 84.3 (13.9)
  Week 52: number analyzed (Participants) | 186 | 85 | 86
  Week 52 | 83.5 (15.5) | 85.1 (13.2) | 82.1 (16.1)

29. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 16
Description: HAQ-DI: participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Week 16
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 19 | 21
Units on a scale | 0.3 (0.4) [lower limit 0.4] | 0.3 (0.4) [lower limit 0.4]

30. Secondary Outcome: Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 24, and 52
Description: as for outcome 29
Time Frame: Week 24 and 52
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
Units on a scale
  Week 24: number analyzed (Participants) | 18 | 8 | 10
  Week 24 | 0.3 (0.4) | 0.2 (0.5) | 0.4 (0.3)
  Week 52: number analyzed (Participants) | 18 | 7 | 10
  Week 52 | 0.3 (0.4) | 0.1 (0.2) | 0.5 (0.3)

31. Secondary Outcome: Patient Global Assessment for Joints on Visual Analog Scale (PJA-VAS) at Week 16
Description: Patient global assessment for joints was measured on a 100 millimeter (mm) VAS scale, where 0 = no pain and 100 = worst possible pain.
Time Frame: Week 16
Population: PP analysis set was used. Here "Number of participants analyzed" signifies participants who were evaluable for this outcome measure at specified category.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 19 | 21
millimeter (mm) | 26.9 (28.3) [lower limit 28.3] | 24.6 (24.3) [lower limit 24.3]

32. Secondary Outcome: Patient Global Assessment for Joints on Visual Analog Scale (PJA-VAS) at Week 24 and 52
Description: as for outcome 31
Time Frame: Week 24 and 52
Population: ETP-PP analysis set was used. Here "Number analyzed" signifies participants who were evaluable for this outcome measure at specified category.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 203 | 95 | 96
mm
  Week 24: number analyzed (Participants) | 18 | 8 | 10
  Week 24 | 29.7 (25.3) | 20.6 (27.1) | 24.9 (20.5)
  Week 52: number analyzed (Participants) | 18 | 7 | 10
  Week 52 | 25.0 (20.3) | 14.7 (16.5) | 29.5 (19.6)

33. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) to Adalimumab at Week 16
Description: Number of participants with treatment emergent Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) to Adalimumab were reported from baseline to week 16. Data was collected using validated bioanalytical method.
Time Frame: Week 16
Population: SAF analysis set was used. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 213 | 202
Participants
  Participants with ADAs | 186 | 179
  Participants with Neutralizing Abs: number analyzed (Participants) | 186 | 179
  Participants with Neutralizing Abs | 70 | 70

34. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs) to Adalimumab at Week 24, 32, 40 and 52
Description: Number of participants With positive treatment emergent Anti-Drug Antibodies (ADAs) and positive Neutralizing Antibodies (NAbs) to Adalimumab were reported. Data was collected using validated bioanalytical method.
Time Frame: Week 24, 32, 40 and 52
Population: ETP-SAF analysis set was used. Here "Number analyzed" signifies participants who were evaluable for this outcome measure at specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 213 | 101 | 101
Participants
  Week 24: ADAs: number analyzed (Participants) | 208 | 96 | 97
  Week 24: ADAs | 185 | 89 | 90
  Week 32: ADAs: number analyzed (Participants) | 200 | 90 | 96
  Week 32: ADAs | 170 | 78 | 85
  Week 40: ADAs: number analyzed (Participants) | 197 | 89 | 92
  Week 40: ADAs | 161 | 72 | 80
  Week 52: ADAs: number analyzed (Participants) | 194 | 87 | 87
  Week 52: ADAs | 162 | 68 | 77
  Week 24: NAb: number analyzed (Participants) | 185 | 89 | 90
  Week 24: NAb | 78 | 42 | 39
  Week 32: NAb: number analyzed (Participants) | 170 | 78 | 85
  Week 32: NAb | 67 | 30 | 32
  Week 40: NAb: number analyzed (Participants) | 160 | 72 | 80
  Week 40: NAb | 70 | 29 | 28
  Week 52: NAb: number analyzed (Participants) | 162 | 68 | 77
  Week 52: NAb | 63 | 29 | 30

35. Secondary Outcome: Anti-Drug Antibodies (ADAs) Titers for Adalimumab at Week 16
Description: Anti-Drug Antibodies (ADAs) Titers for adalimumab at week 16 was reported. Data was collected using validated bioanalytical method.
Time Frame: Week 16
Population: SAF analysis set was used. Here "Number of Participants analyzed" signifies those who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Titers
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 213 | 202
Titers | 8.0 (1) [1 to 2048] | 8.0 (1) [1 to 1024]

36. Secondary Outcome: Anti-Drug Antibodies (ADAs) Titers for Adalimumab at Week 24, 32, 40 and 52
Description: Anti-Drug Antibodies (ADAs) Titers for adalimumab at Week 24, 32, 40 and 50 was reported. Data was collected using validated bioanalytical method.
Time Frame: Week 24, 32, 40 and 52
Population: ETP-SAF analysis set was used. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified category.
Measure: Median (Full Range); unit: Titers
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 213 | 101 | 101
Titers
  Week 24: number analyzed (Participants) | 185 | 89 | 90
  Week 24 | 16.0 [1 to 4096] | 16.0 [1 to 4096] | 16.0 [1 to 4096]
  Week 32: number analyzed (Participants) | 170 | 78 | 85
  Week 32 | 16.0 [1 to 1024] | 16.0 [1 to 8192] | 16.0 [1 to 16384]
  Week 40: number analyzed (Participants) | 161 | 72 | 80
  Week 40 | 16.0 [1 to 8192] | 16.0 [1 to 8192] | 16.0 [1 to 16384]
  Week 52: number analyzed (Participants) | 162 | 68 | 77
  Week 52 | 8.0 [1 to 4096] | 16.0 [1 to 4096] | 8.0 [1 to 4096]

37. Secondary Outcome: Observed Serum Concentration at Week 16
Description: Observed serum concentrations at week 16 were reported.
Time Frame: Week 16
Population: The Pharmacokinetic (PK) Analysis Set included all participants in the SAF who also had at least 1 measurable post-dose concentration. Here "Number of Participants analyzed" signifies those who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira
Number analyzed (Participants) | 192 | 170
Nanogram per milliliter (ng/mL) | 6990 (4504) [lower limit 4504] | 6410 (4152) [lower limit 4152]

38. Secondary Outcome: Observed Serum Concentration at Week 24 and 52
Description: Observed serum concentrations at week 24 and 52 were reported.
Time Frame: Week 24 and 52
Population: The ETP-PK analysis included all participants in ETP SAF who had at least 1 measurable post-dose concentration in ETP, without any important protocol deviations that could have impacted quality of PK data during ETP. Here "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
Number analyzed (Participants) | 198 | 87 | 92
ng/mL
  Week 24: number analyzed (Participants) | 184 | 86 | 85
  Week 24 | 6240 (4569) | 5870 (4516) | 6430 (4610)
  Week 52: number analyzed (Participants) | 161 | 76 | 72
  Week 52 | 6910 (5750) | 5930 (4529) | 6600 (5394)

ADVERSE EVENTS:
Time Frame: Core Treatment period: Baseline up to Week 16; Extended Treatment Period: Baseline up to Week 54
Arm/Group | MSB11022 (Core Treatment Period) | EU-Humira | MSB11022 (Extended Treatment Period) | EU-Humira/EU-Humira | EU-Humira/MSB11022
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/220 | 0/213 | 1/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 8/221 | 6/220 | 12/213 | 3/101 | 4/101
Other Adverse Events (participants affected / at risk) | 30/221 | 34/220 | 59/213 | 32/101 | 25/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSB11022 (Core Treatment Period) (N=221) | EU-Humira (N=220) | MSB11022 (Extended Treatment Period) (N=213) | EU-Humira/EU-Humira (N=101) | EU-Humira/MSB11022 (N=101)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival cyst (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular compression (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MSB11022 (Core Treatment Period) (N=221) | EU-Humira (N=220) | MSB11022 (Extended Treatment Period) (N=213) | EU-Humira/EU-Humira (N=101) | EU-Humira/MSB11022 (N=101)
Injection site erythema (General disorders) | 11 (18) | 13 (19) | 9 (19) | 5 (25) | 6 (31)
Injection site pain (General disorders) | 11 (52) | 11 (28) | 12 (54) | 4 (4) | 5 (18)
Nasopharyngitis (Infections and infestations) | 13 (13) | 15 (16) | 31 (36) | 12 (14) | 16 (16)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 11 (15) | 5 (7) | 4 (4)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 11 (12) | 10 (11) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other